CLINICAL TRIAL: NCT01666613
Title: A Phase I, Single-centre, Open-label, Partly Randomised, Cross-over Single Dose Study in Healthy Volunteers to Evaluate the Absolute Pulmonary Bioavailability of AZD8683 When Administered Inhaled Via a New Dry Powder Inhaler and Via Turbuhaler™
Brief Title: A Study in Healthy Subjects to Investigate Pharmacokinetics of AZD8683 When Administered in Different Ways
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1883C00008; EudraCT number 2012-002901-23
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Phase I, Healthy volunteers, pharmacokinetics; Bioavailability; AUC

ARMS (4):
- 1 (Experimental): AZD8683 iv
  Interventions: Drug: AZD8683
- 2 (Experimental): AZD8683 oral
  Interventions: Drug: AZD8683
- 3 (Experimental): AZD8683 inhalation New Dry Powder Inhaler
  Interventions: Drug: AZD8683
- 4 (Experimental): AZD8683 inhalation Turbuhaler™
  Interventions: Drug: AZD8683

INTERVENTIONS:
Drug: AZD8683 — Solution for injection, administered as intravenous infusion Total dose of 100µg AZD8683
  Arms: 1
Drug: AZD8683 — Solution to be administered orally Total dose of 950 µg AZD8683
  Arms: 2
Drug: AZD8683 — Dry powder inhaled via New Dry Powder Inhaler, 540 µg delivered dose AZD8683
  Arms: 3
Drug: AZD8683 — Dry powder inhaled via Turbuhaler™, 600 µg delivered dose AZD8683
  Arms: 4

SUMMARY:
The purpose of this study is to look at drug levels of AZD8683 in blood when the drug is administered in different ways - orally, intravenously or inhaled (with two different devices), to healthy subjects

DETAILED DESCRIPTION:
A Phase I, Single-centre, Open-label, Partly Randomised, Cross-over Single Dose Study in Healthy Volunteers to Evaluate the Absolute Pulmonary Bioavailability of AZD8683 when Administered Inhaled via a New Dry Powder Inhaler and via Turbuhaler™

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or women of non-childbearing potential aged 18-45 years inclusive with suitable veins for cannulation or repeated vein puncture
* Have a body mass index (BMI) between 19 and 30 kg/m2 (inclusive) and weight between 50 and 100 kg (inclusive)
* Be able to inhale from the inhaler devices used in the study.

Exclusion Criteria:

* History of any clinically significant disease or disorder
* Current smokers
* Any clinically relevant abnormal findings in physical examination or laboratory values.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Absolute pulmonary bioavailability of AZD8683 delivered by the new dry powder inhaler in terms of: Fpulmonary | Blood samples taken pre-dose and at 5, 15 and 30 minutes and 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post dose.

SECONDARY OUTCOMES:
Absolute pulmonary bioavailability of AZD8683 delivered by the Turbuhaler™ in terms of: Fpulmonary | Blood samples taken pre-dose and at 5, 15 and 30 minutes and 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post dose.
Pharmacokinetics of AZD8683 following administration in terms of oral inhalation by Turbuhaler™ and New Dry Powder Inhaler in terms of: Finhalation total, FrelAUC, Frel Cmax and Foral | Blood samples taken pre-dose and at 5, 15 and 30 minutes and 1, 2, 4, 8, 12,24, 36, 48, 72, 96, 120 and 144 hours post dose.
Pharmacokinetics of AZD8683 following oral administration in terms of: Fpo | Blood samples taken pre-dose and at 5, 15 and 30 minutes and 1, 2, 4, 8, 12 ,24, 36, and 48 hours post dose.
Pharmacokinetics of AZD8683 following oral administration and oral inhalation by Turbuhaler™ and New Dry Powder inhaler in terms of : AUC, AUC(0-t), Cmax, tmax, t½λz, MRT and MAT. | Blood samples taken pre-dose and at 5, 15 and 30 minutes and 1, 2, 4, 8, 12,24, 36, 48, 72 96, 120 and 144 hours post dose.
Pharmacokinetics of AZD8683 following i.v. administration in terms of: CL, Vz, and Vss | Blood samples taken pre-dose and at 5, 15, 20, 25 and 40 minutes and 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 and 144 hours post dose.
Safety profile in terms of adverse events, ECG, heart rate, blood pressure, body temperature, physical examination, spirometry, haematology, clinical chemistry and urinalysis. | Screening to 4 weeks after last dose.
  No formal statistical tests will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, MD, Study Director — AstraZeneca R&D, Molndal Sweden